CLINICAL TRIAL: NCT01235247
Title: Electronic Medical Records to Improve Patient & Public Health in Rural Kenya
Brief Title: Decision Support AMPATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indiana University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Moi Teaching and Referral Hospital (Other)
Responsible Party: William M. Tierney, MD, Indiana University School of Medicine
Purpose: Health Services Research
Other Study IDs: 0709-63
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2007-09

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- reminders, no reminder (Experimental)
  Interventions: Behavioral: reminders vs. no reminders

INTERVENTIONS:
Behavioral: reminders vs. no reminders — Intervention providers will receive clinical reminders as part of patient care, and control group providers will not receive the reminders

SUMMARY:
Computer-generated clinical reminders offered to providers will improve compliance with care guidelines and impact outcomes in resource-limited clinics.

DETAILED DESCRIPTION:
The investigators will assess the effects of computer-generated reminders for the 3 cohorts of patients: (1) pregnant women; (2) HIV-exposed infants; and (3) adults and children co-infected with TB and HIV identified from the AMPATH clinics. Patients will be randomized to either receive the reminders as part of a paper summary, or to not have any of the reminders in their summary. Reminders implemented will vary by type of patient population. Comparisons will be made between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women, children born to HIV+ mothers, and TB/HIV co-infected patients visiting these clinics during the this study will be included.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2011-02; Primary Completion 2011-10 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Compliance rates with care guidelines | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- USAID-AMPATH Clinics, Eldoret, Kenya

REFERENCES:
- [Derived] Were MC, Nyandiko WM, Huang KT, Slaven JE, Shen C, Tierney WM, Vreeman RC. Computer-generated reminders and quality of pediatric HIV care in a resource-limited setting. Pediatrics. 2013 Mar;131(3):e789-96. doi: 10.1542/peds.2012-2072. Epub 2013 Feb 25. PMID 23439898